CLINICAL TRIAL: NCT02561403
Title: Cognitive Reserve and Training in Older Veterans With Traumatic Brain Injury: Study 2
Brief Title: Brain Aging in Veterans (BRAVE) Training: A Cognitive Training Pilot Trial in Older Veterans With Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Allison Kaup, Clinical Research Psychologist, San Francisco Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 14-14955
Record Dates: First submitted 2015-09-23; First posted 2015-09-28 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: traumatic brain injury (TBI); aging; cognitive training; Cognitive Aging
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- EVO multitask video game (Experimental)
  Interventions: Behavioral: EVO multitask video game
- EVO words video game (Experimental)
  Interventions: Behavioral: EVO words video game
- Assessment Only (No Intervention)

INTERVENTIONS:
Behavioral: EVO multitask video game — Participants will play a multitasking game for 4 weeks
  Arms: EVO multitask video game
Behavioral: EVO words video game — Participants will play a word puzzle game for 4 weeks
  Arms: EVO words video game

SUMMARY:
The purpose of this study is to conduct a pilot trial investigating cognitive training in older Veterans with a history of traumatic brain injury (TBI) to assess training effects, acceptability of training to participants, and to explore whether other factors influence training effects.

DETAILED DESCRIPTION:
A study of older Veterans (60-85 years old) who have 1) a history of repetitive mild TBI or at least one moderate TBI and 2) subjective cognitive complaints. Participants will be randomized to one of three conditions for 4 weeks: Project:Evolution (EVO) multitask video game, EVO words video game, or an assessment only control condition. Participants will complete assessment visits at baseline, post-intervention (1 month after baseline), and 3 months post-intervention (4 months after baseline).

ELIGIBILITY:
Inclusion Criteria:

1. Ages 60-85
2. Have experienced more than one mild TBI or at least one moderate TBI over their lifetime
3. Have current cognitive problems based on self-report
4. Vision adequate to see test stimuli
5. Hearing adequate to understand the examiner
6. Fluent in English in order to understand task instructions
7. Demonstrate capacity to consent to participate in research
8. Mini-Mental Status Exam (MMSE) score ≥ 25

Exclusion Criteria:

1. History of penetrating brain injury
2. Active disabling neurological condition (e.g., stroke, brain tumor, multiple sclerosis)
3. History of severe psychiatric illness (i.e., schizophrenia, bipolar disorder, schizoaffective disorder)
4. Active drug use or active heavy alcohol use
5. History of severe TBI
6. History of a dementia diagnosis
7. Individuals who are physically unable to use an iPad for 30 minutes at a time per day will be excluded, such as individuals with debilitating arthritis or tremor

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Acceptability based on participant ratings | Acceptability ratings assessed post-intervention (1-month after baseline)
Participant adherence to game play | Total adherence over the 4 week intervention phase
Change in cognitive functioning based on neurocognitive test battery | Baseline, post-intervention (1-month after baseline), and 3-months post-intervention (4-months after baseline)

SECONDARY OUTCOMES:
Change in self-reported everyday cognitive functioning [Neuro-QOL (Quality of Life in Neurological Disorders) Cognitive Function inventory] | Baseline, post-intervention (1-month after baseline), and 3-months post-intervention (4-months after baseline)
Change in everyday functioning [University of California San Diego (UCSD) Performance Based Skills Assessment (UPSA)] | Baseline, post-intervention (1-month after baseline), and 3-months post-intervention (4-months after baseline)
Change in mood symptoms (Geriatric Depression Scale) | Baseline, post-intervention (1-month after baseline), and 3-months post-intervention (4-months after baseline)
Change in EVO performance (EVO Monitor) | Baseline, post-intervention (1-month after baseline), and 3-months post-intervention (4-months after baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kaup, PhD, Principal Investigator — San Francisco Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, California
  - Veterans Home of California, Yountville, California